CLINICAL TRIAL: NCT00065845
Title: CARE: A Randomized Trial of Colpopexy and Urinary Reduction Efforts
Brief Title: Colpopexy and Urinary Reduction Efforts (CARE) Protocol
Acronym: CARE
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Susan Meikle, MD, NICHD
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: U01HD041249 (NIH); U10HD041268 (NIH); U10HD041248 (NIH); U10HD041250 (NIH); U10HD041261 (NIH); U10HD041263 (NIH); U10HD041269 (NIH); U10HD041267 (NIH)
Record Dates: First submitted 2003-08-01; First posted 2003-08-05 (Estimated); Last update posted 2011-01-11 (Estimated); Status verified 2010-10

CONDITIONS: Urinary Incontinence, Stress; Uterine Prolapse; Vaginal Prolapse
Keywords: Urinary incontinence; Pelvic organ prolapse; Stress incontinence; Sacrocolpopexy; Burch urethropexy; Surgical Trials
MeSH Terms: conditions — Urinary Incontinence, Stress; Uterine Prolapse; Urinary Incontinence; Pelvic Organ Prolapse

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Abdominal Sacral Colpopexy with no Burch colposuspension (No Intervention): Abdominal sacral colpopexy is performed through a laparotomy approach.
- Abdominal Sacral Colpopexy with Burch Colposuspension (Experimental): The Burch colposuspension procedure entails the retropubic placement of at least two stitches in the vaginal tissue lateral to each side of the urethra, and suspension of these stitches from Cooper's ligament (the iliopectineal line at the superior aspect of the posterior pubic bone).
  Interventions: Procedure: Burch urethropexy at time of sacrocolpopexy

INTERVENTIONS:
Procedure: Burch urethropexy at time of sacrocolpopexy — The Burch colposuspension procedure entails the retropubic placement of at least two stitches in the vaginal tissue lateral to each side of the urethra, and suspension of these stitches from Cooper's ligament (the iliopectineal line at the superior aspect of the posterior pubic bone).
  Arms: Abdominal Sacral Colpopexy with Burch Colposuspension

SUMMARY:
Pelvic organ prolapse occurs when the muscles holding pelvic organs (e.g., the uterus or bladder) weaken and the organs fall or slide down into the vagina. Pelvic organ prolapse can be corrected with surgery. However, women who have this surgery may develop urinary incontinence. This study will determine how doctors can predict this problem and whether an additional surgical procedure at the time of prolapse surgery can prevent the development of urinary incontinence.

DETAILED DESCRIPTION:
Many women have surgery for pelvic organ prolapse (cystocele, uterine prolapse, rectocele). Women with advanced pelvic organ prolapse may experience stress urinary incontinence following surgery to repair the prolapse. Development of incontinence is unpredictable. This study will determine which, if any, clinical tests are useful for predicting post-operative urinary incontinence. The study will also determine if a Burch urethropexy should be performed routinely or selectively at the time of sacrocolpopexy in continent women.

Women with pelvic organ prolapse who are scheduled for prolapse repair will be randomized to a Burch urethropexy group or to a control group. Women in the Burch group will undergo urethropexy at the time of prolapse repair. Assessments will include a quality of life telephone interview, urodynamic testing, and physical examination. Follow-up evaluations occur at 6 weeks, 3 months, and 1 and 2 years following surgery. Post-operative phone interviews will occur at 3 months, 6 months, and 1 and 2 years.

ELIGIBILITY:
Inclusion Criteria

1. Eligibility for primary procedure (sacrocolpopexy)
2. Eligibility for secondary procedure (Burch colposuspension)
3. Stage II-IV anterior vaginal prolapse, defined as POP-Q Point Aa at -1, 0, +1, +2, or +3 cm.
4. Negative stress incontinence screen
5. Negative stress incontinence screen (MESA questionnaire)

Exclusion Criteria

1. Contraindication for sacrocolpopexy or Burch colposuspension.

   * Anatomic contraindication for Burch colposuspension (i.e., Point Aa fixed at -2 or -3 cm).
   * Surgeon judgment that a contraindication to Burch colposuspension exists.
2. Anticipated geographic relocation within the first three months after surgery (e.g., within approximately 6 months of screening).
3. Inability to provide informed consent or to complete testing or data collection.
4. Currently pregnant.

Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2002-04; Primary Completion 2007-03 (Actual); Study Completion 2007-04 (Actual)

PRIMARY OUTCOMES:
Stress urinary continence | 3 months
  Patients will be categorized as stress continent or stress incontinent on the basis of symptom assessment and stress testing. The symptoms will be assessed by the stress incontinence subscale of the Pelvic Floor Distress Inventory (PFDI).

SECONDARY OUTCOMES:
Complications at surgery | 2 years
  Complications at surgery
Occurrence of other lower urinary tract symptoms | 3 mo, 2 years
  measured by the urgency and obstructed voiding subscales of the PFDI
Other pelvic symptoms and health-related quality of life | 3 mo, 2 years
  includes bowel function and sexual function

CONTACTS AND LOCATIONS:
Overall Officials: Linda Brubaker, MD, Principal Investigator — Loyola University
Locations (7):
- United States (7):
  - The University of Alabama at Birmingham, Birmingham, Alabama
  - Loyola University Medical Center, Maywood, Illinois
  - University of Iowa College of Medicine, Iowa City, Iowa
  - Johns Hopkins School of Medicine, Baltimore, Maryland
  - University of North Carolina at Chapel Hill, Chapel Hill, North Carolina
  - Magee-Womens Hospital, Pittsburgh, Pennsylvania
  - Baylor College of Medicine, Houston, Texas

REFERENCES:
- [Result] Brubaker L, Cundiff GW, Fine P, Nygaard I, Richter HE, Visco AG, Zyczynski H, Brown MB, Weber AM; Pelvic Floor Disorders Network. Abdominal sacrocolpopexy with Burch colposuspension to reduce urinary stress incontinence. N Engl J Med. 2006 Apr 13;354(15):1557-66. doi: 10.1056/NEJMoa054208. PMID 16611949
- [Result] Burgio KL, Nygaard IE, Richter HE, Brubaker L, Gutman RE, Leng W, Wei J, Weber AM; Pelvic Floor Disorders Network. Bladder symptoms 1 year after abdominal sacrocolpopexy with and without Burch colposuspension in women without preoperative stress incontinence symptoms. Am J Obstet Gynecol. 2007 Dec;197(6):647.e1-6. doi: 10.1016/j.ajog.2007.08.048. PMID 18060965
- [Result] Bradley CS, Nygaard IE, Brown MB, Gutman RE, Kenton KS, Whitehead WE, Goode PS, Wren PA, Ghetti C, Weber AM; Pelvic Floor Disorders Network. Bowel symptoms in women 1 year after sacrocolpopexy. Am J Obstet Gynecol. 2007 Dec;197(6):642.e1-8. doi: 10.1016/j.ajog.2007.08.023. PMID 18060963
- [Result] Visco AG, Brubaker L, Nygaard I, Richter HE, Cundiff G, Fine P, Zyczynski H, Brown MB, Weber AM; Pelvic Floor Disorders Network. The role of preoperative urodynamic testing in stress-continent women undergoing sacrocolpopexy: the Colpopexy and Urinary Reduction Efforts (CARE) randomized surgical trial. Int Urogynecol J Pelvic Floor Dysfunct. 2008 May;19(5):607-14. doi: 10.1007/s00192-007-0498-2. Epub 2008 Jan 9. PMID 18185903
- [Result] Nygaard I, Handa VL, Brubaker L, Borello-France D, Wei J, Wells E, Goode P; Pelvic Floor Disorders Network. Changes in physical activity after abdominal sacrocolpopexy for advanced pelvic organ prolapse. Am J Obstet Gynecol. 2008 May;198(5):570.e1-5. doi: 10.1016/j.ajog.2008.01.044. PMID 18455536
- [Result] Wren PA, Janz NK, FitzGerald MP, Barber MD, Burgio KL, Cundiff GW, Nygaard IE, Zyczynski HM, Gao X; Pelvic Floor Disorders Network. Optimism in women undergoing abdominal sacrocolpopexy for pelvic organ prolapse. J Am Coll Surg. 2008 Aug;207(2):240-5. doi: 10.1016/j.jamcollsurg.2008.02.019. Epub 2008 May 12. PMID 18656053
- [Result] Goode PS, Fitzgerald MP, Richter HE, Whitehead WE, Nygaard I, Wren PA, Zyczynski HM, Cundiff G, Menefee S, Senka JM, Gao X, Weber AM; Pelvic Floor Disorders Network. Enhancing participation of older women in surgical trials. J Am Coll Surg. 2008 Sep;207(3):303-11. doi: 10.1016/j.jamcollsurg.2008.03.012. Epub 2008 May 19. PMID 18722933
- [Result] Brubaker L, Nygaard I, Richter HE, Visco A, Weber AM, Cundiff GW, Fine P, Ghetti C, Brown MB. Two-year outcomes after sacrocolpopexy with and without burch to prevent stress urinary incontinence. Obstet Gynecol. 2008 Jul;112(1):49-55. doi: 10.1097/AOG.0b013e3181778d2a. PMID 18591307
- [Result] Cundiff GW, Varner E, Visco AG, Zyczynski HM, Nager CW, Norton PA, Schaffer J, Brown MB, Brubaker L; Pelvic Floor Disorders Network. Risk factors for mesh/suture erosion following sacral colpopexy. Am J Obstet Gynecol. 2008 Dec;199(6):688.e1-5. doi: 10.1016/j.ajog.2008.07.029. Epub 2008 Oct 31. PMID 18976976
- [Result] Bradley CS, Kenton KS, Richter HE, Gao X, Zyczynski HM, Weber AM, Nygaard IE; Pelvic Floor Disorders Network. Obesity and outcomes after sacrocolpopexy. Am J Obstet Gynecol. 2008 Dec;199(6):690.e1-8. doi: 10.1016/j.ajog.2008.07.030. Epub 2008 Oct 9. PMID 18845288
- [Result] Barber MD, Brubaker L, Nygaard I, Wheeler TL 2nd, Schaffer J, Chen Z, Spino C; Pelvic Floor Disorders Network. Defining success after surgery for pelvic organ prolapse. Obstet Gynecol. 2009 Sep;114(3):600-609. doi: 10.1097/AOG.0b013e3181b2b1ae. PMID 19701041
- [Derived] Lukacz ES, Sridhar A, Chermansky CJ, Rahn DD, Harvie HS, Gantz MG, Varner RE, Korbly NB, Mazloomdoost D; Eunice Kennedy Shriver National Institute of Child Health and Human Development Pelvic Floor Disorders Network (PFDN). Sexual Activity and Dyspareunia 1 Year After Surgical Repair of Pelvic Organ Prolapse. Obstet Gynecol. 2020 Sep;136(3):492-500. doi: 10.1097/AOG.0000000000003992. PMID 32769645
- [Derived] Barber MD, Chen Z, Lukacz E, Markland A, Wai C, Brubaker L, Nygaard I, Weidner A, Janz NK, Spino C. Further validation of the short form versions of the Pelvic Floor Distress Inventory (PFDI) and Pelvic Floor Impact Questionnaire (PFIQ). Neurourol Urodyn. 2011 Apr;30(4):541-6. doi: 10.1002/nau.20934. Epub 2011 Feb 22. PMID 21344495